CLINICAL TRIAL: NCT04599634
Title: A Phase 1 Study of Venetoclax With Obinutuzumab and Magrolimab (VENOM) in Relapsed and Refractory Indolent B-cell Malignancies
Brief Title: Venetoclax With Obinutuzumab and Magrolimab (VENOM) in Relapsed and Refractory Indolent B-cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Roschewski, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200162; 20-C-0162
Record Dates: First submitted 2020-10-22; First posted 2020-10-23 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma; Chronic Lymphocytic Lymphoma; B-Cell Lymphoma
Keywords: CD47; Monoclonal Anti-CD20 Antibody; Follicular Lymphoma; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Lymphoma, B-Cell | interventions — obinutuzumab; venetoclax; magrolimab; Acetaminophen; Diphenhydramine; Prednisone; Prednisolone; Methylprednisolone; Methylprednisolone Hemisuccinate; Methylprednisolone Acetate; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Experimental treatment: FL dose expansion (Experimental): Window of magrolimab intravenous (IV) with a 1 mg/kg priming dose followed by 30mg/kg loading and maintenance doses + obinutuzumab IV 1000mg combination for two (2) cycles (28-days each, Cycles -2 and -1), then venetoclax will be added at target dose (dose determined from Arm 1). Triplet combination treatment with magrolimab + obinutuzumab + venetoclax will be 6 cycles (28-days each, Cycles 1-6); further treatment will be response-adapted.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax; Drug: Magrolimab; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Prednisone/prednisolone; Drug: Methylprednisolone; Diagnostic Test: CT Scan chest/abdomen/pelvis; Diagnostic Test: MRI; Diagnostic Test: 18-FDG-PET; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration
- Experimental treatment: FL Dose-finding (Experimental): Magrolimab intravenous (IV) with a 1 mg/kg priming dose followed by 30mg/kg loading and maintenance doses + obinutuzumab IV 1000mg + venetoclax 800mg by mouth (PO) combination administered to 6 patients for six (6) cycles (28-days each, Cycles 1-6); further treatment with additional cycles will be response-adapted. Note: Dose-limiting toxicity (DLT) assessment of the magrolimab + obinutuzumab + venetoclax triplet will take place during Cycle 1. If =2 patients experience DLT, an additional 6 patients will be enrolled at Dose level (DL (-1) of venetoclax 600mg with magrolimab and obinutuzumab.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax; Drug: Magrolimab; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Prednisone/prednisolone; Drug: Methylprednisolone; Diagnostic Test: CT Scan chest/abdomen/pelvis; Diagnostic Test: MRI; Diagnostic Test: 18-FDG-PET; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration
- Experimental treatment: MZL, MCL, and CLL Dose-finding (Experimental): Magrolimab intravenous (IV) with a 1 mg/kg priming dose followed by 30mg/kg loading and maintenance doses + obinutuzumab IV 1000mg + venetoclax ramp-up to target dose of 400mg over 5 weeks (35 days, Cycle 1) administered to 6 patients. Triplet combination of magrolimab + obinutuzumab + venetoclax (target dose, no ramp-up) will continue for five (5) additional cycles (28-days each, Cycles 2-6); further treatment with additional cycles will be response-adapted. Note: Dose-limiting toxicity (DLT) assessment of the magrolimab + obinutuzumab + venetoclax triplet will take place during Cycle 1. If =2 patients experience DLT, an additional 6 patients will be enrolled at Dose level (DL (-1) of venetoclax 200mg with magrolimab and obinutuzumab.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax; Drug: Magrolimab; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Prednisone/prednisolone; Drug: Methylprednisolone; Diagnostic Test: CT Scan chest/abdomen/pelvis; Diagnostic Test: MRI; Diagnostic Test: 18-FDG-PET; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration
- Experimental treatment: mzl, MCL, CLL dose expansion (Experimental): Window of magrolimab intravenous (IV) with a 1 mg/kg priming dose followed by 30mg/kg loading and maintenance doses + obinutuzumab IV 1000mg combination for two (2) cycles (28-day cycles, Cycles -2 and -1), then venetoclax safety ramp-up to target dose (dose determined from Arm 2) over 5 weeks (35-days, Cycle 1). Triplet combination treatment with magrolimab + obinutuzumab + venetoclax (target dose, no ramp-up) will continue for 5 additional cycles (28-days each, Cycles 2-6); further treatment will be response-adapted.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax; Drug: Magrolimab; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Prednisone/prednisolone; Drug: Methylprednisolone; Diagnostic Test: CT Scan chest/abdomen/pelvis; Diagnostic Test: MRI; Diagnostic Test: 18-FDG-PET; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration

INTERVENTIONS:
Drug: Obinutuzumab — Administered intravenously, on Days 1, 2, 8 and 15 of Cycle 1 at doses escalating from 100mg - 1000mg then on the first day for all subsequent cycles at 1000mg for dose finding phase. For expansion phase, administered on Days 1, 2, 8 and 15 of Cycle 2 at doses escalating from 100mg - 1000mg then on the first day for all subsequent cycles at 1000mg.
  Other Names: Gazyna; Afutuzumab; GA101
Drug: Venetoclax — For follicular lymphoma (FL) patients in dose finding phase, administered orally at a dose of 600mg or 800mg depending on tolerance, daily, cycles 1-12. For MZL (Marginal Zone Lymphoma), MCL (Mantle Cell Lymphoma) or CLL (Chronic Lymphocytic Leukemia) patients in dose finding phase administered at an escalating dose from 20mg-400mg Cycle 1 on days 1-35, and at a dose of 400mg per day for Cycles 2-12. Patients in expansion phase will receive target dose established from dose finding cohorts daily for all 12 cycles.
  Other Names: GDC-0199; ABT-199; RG-7601
Drug: Magrolimab — Administered intravenously, starting at 1 mg/kg on second day of first cycle then 30mg/kg on days 8, 15 and 22 of cycle 1 and days 1 and 15 of cycles 2-12 for patients in both the dose finding and expansion phases.
  Other Names: 5F9; GS-4721; ONO-7913
Drug: Acetaminophen — Premedication with 650mg acetaminophen 30-60 minutes prior to obinutuzumab doses.
  Other Names: Tylenol; Ofirmev; FeverAll
Drug: Diphenhydramine — Premedication with 25-50mg diphenhydramine 30-60 minutes prior to obinutuzumab doses.
  Other Names: Benadryl; Banophen; Nytol
Drug: Prednisone/prednisolone — Premedication with 100mg intravenous prednisone/prednisolone 30-60 minutes before obinutuzumab infusion.
  Other Names: Rayos; Deltasone; Prednisone Intensol
Drug: Methylprednisolone — Premedication with intravenous methylprednisolone 80mg 30-60 minutes before obinutuzumab infusion.
  Other Names: Solu-Medrol; Depo-Medrol; Medrol
Diagnostic Test: CT Scan chest/abdomen/pelvis — Screening, baseline, window Cycle -1/pre cycle 1, cycles 6-12; cycles 3-9, end of treatment and follow-up.
  Other Names: Computed tomography scan chest/abdomen/pelvis
Diagnostic Test: MRI — Screening, baseline, window Cycle -1/pre cycle 1, cycles 6-12; cycles 3-9, end of treatment and follow-up.
  Other Names: Magnetic resonance imaging
Diagnostic Test: 18-FDG-PET — Baseline, Cycle -1, Day 1, window Cycle -1/pre cycle 1, cycles 6-12, end of treatment and follow-up.
  Other Names: 18F-fluorodeoxyglucose positron emission tomography
Procedure: Bone Marrow Biopsy — Screening, Cycle 7-12, Day 1 and end of treatment.
  Other Names: BM Bx
Procedure: Bone Marrow Aspiration — Screening, Cycle 7-12, Day 1 and end of treatment.
  Other Names: BM aspiration

SUMMARY:
Background:

B-cell lymphoma is a cancer of certain white blood cells (called lymphocytes). These cells are found in lymph nodes. The cancer can cause enlargement of the lymph nodes leading to pain and discomfort. Swollen lymph nodes can also press on nearby organs such as liver and kidneys which can affect normal functioning of the organs. Researchers think that a new combination of drugs may be able to help.

Objective:

To find out if it is safe to give the combination of Magrolimab, Obinutuzumab and Venetoclax to people with B-cell lymphomas.

Eligibility:

Adults age 18 and older with an indolent B-cell lymphoma whose disease has returned or progressed after other treatment. Indolent B-cell lymphoma for this protocol is defined as having either follicular lymphoma, mantle cell lymphoma, chronic lymphocytic leukemia/small lymphocytic lymphoma or marginal zone lymphoma.

Design:

Participants will be screened under a separate protocol.

Participants will have 28-day 'cycles' of treatment. They will take Venetoclax by mouth daily. They will get Obinutuzumab and Magrolimab by intravenous (IV) infusion. Treatment will last for about 8 months. They may be able to have more cycles of treatment if their cancer is responding well.

Participants will have physical exams, medical histories, and medicine reviews. Data about how they function in their daily activities will be obtained. They will have blood and urine tests. They may have bone marrow tests.

Participants will have imaging scans. These will include computed tomography (CT) and/or magnetic resonance imaging (MRI) scans and positron emission tomography (PET) scans.

Participants may give a cheek swab or saliva sample. They may give tumor tissue and bone marrow samples. These samples may be used for gene testing.

Participants will have a follow-up visit about 30 days after treatment ends. Then they will have visits every 3 months for the first 2 years, every 6 months for the next 3 years, and then yearly after that.

DETAILED DESCRIPTION:
Background:

* Indolent B-cell malignancies are associated with frequent disease relapse
* Standard frontline therapy includes a monoclonal anti-cluster of differentiation 20 (CD20) antibody with or without chemotherapy; novel targeted therapies have changed the treatment landscape and are preferred therapy for some patients with high-risk molecular features
* Targeted therapies given indefinitely add to drug resistance, treatment-emergent toxicities, and non-compliance
* Cluster of differentiation 47 (CD47) is a rational target for indolent B-cell malignancies; CD47 expression is higher in tumor cells than normal B-cells, and blocking CD47 results in phagocytosis of tumor cells
* Magrolimab is an anti-CD47 monoclonal antibody with activity in refractory indolent lymphomas when combined with rituximab (a first generation anti-CD20 monoclonal antibody)
* Obinutuzumab is a novel anti-CD20 monoclonal antibody with enhanced binding to the Fc receptor that may improve antibody-dependent cell-mediated cytotoxicity (ADCC), and phagocytosis, when combined with magrolimab
* We aim to test the safety and efficacy of venetoclax when added to the backbone of magrolimab and obinutuzumab in patients with relapsed or refractory indolent B-cell malignancies
* Treatment duration will be response-adapted and time-limited in all patients

Objective:

-To determine the safety of the triplet combination of venetoclax, magrolimab and obinutuzumab in relapsed and refractory indolent B-cell malignancies

Eligibility:

* Follicular lymphoma (FL) (grades 1-2, or 3a), marginal zone lymphoma (MZL), mantle cell lymphoma (MCL) or chronic lymphocytic leukemia (CLL) with greater than or equal to 2 prior therapies, with at least one of those therapies containing an anti-CD20 monoclonal antibody
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate bone marrow and organ function

Design:

* Phase 1 study with expansion cohorts of up to 76 patients with relapsed or refractory FL, MZL, MCL or CLL
* The safety profile of magrolimab, venetoclax, and obinutuzumab will first be determined in a dose-finding phase of up to 24 patients (6-12 patients with FL and 6-12 patients with MZL, MCL or CLL). Patients without dose-limiting toxicity (DLT) will receive an additional 5 cycles (total 6 cycles) of the triplet combination.
* After dose-finding is completed, expansion cohorts of each histology will first receive magrolimab and obinutuzumab for 2 cycles in a window for translational research. After the window, venetoclax will be added and patients will receive 6 cycles (total 8 cycles) of the triplet combination.
* Patients who achieve a complete response (CR) (after a total of 6 cycles of the triplet combination) will stop treatment and initiate active monitoring with radiologic imaging and assays for circulating tumor DNA (ctDNA); if these patients relapse, they can be retreated with 6 additional cycles. Patients who achieve partial response (PR) after 6 cycles of the triplet will continue for an additional 6 cycles; then, will initiate active monitoring.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have a confirmed histologic diagnosis of an indolent cluster of differentiation 20 (CD20) positive B-cell lymphoma according to the criteria established by the 2016 version of the World Health Organization (WHO) classification system. Lymphomas with any prior CD20 expression (by immunohistochemistry or flow cytometry) will be considered eligible. Diagnosis must be confirmed by Laboratory of Pathology, National Cancer Institute (NCI) and the following indolent B-cell lymphomas are included:

  * Follicular lymphoma (FL): must be grade 1-2 or 3a
  * Marginal zone lymphoma (MZL)
  * Mantle cell lymphoma (MCL)
  * Chronic lymphocytic leukemia (CLL)
* Participant must have relapsed and/or refractory disease, as defined below:
* FL: relapsed after and/or refractory to at least two (2) prior lines of therapy with at least one of those therapies containing an anti-CD20 monoclonal antibody.

NOTE: Participants with FL may be eligible after one (1) prior line of therapy if they have either:

* Follicular lymphoma international prognostic index (FLIPI) >=2 (120)
* Disease progression within 24 months of the end of last therapy (POD24)
* MZL: relapsed after and/or refractory to at least two (2) prior lines of therapy, with at least one containing an anti-CD20 monoclonal antibody.
* MCL: relapsed after and/or refractory to at least two (2) prior lines of therapy, with at least one containing an anti-CD20 monoclonal antibody.

NOTE: Participants with MCL may be eligible after one (1) prior line of therapy if they have either:

* Blastoid or pleomorphic histology
* 17p deletion
* Tumor protein p53 (TP53) mutation or deletion
* Antigen Kiel 67 (Ki67) >=30%
* Received a Bruton tyrosine kinase (BTK) inhibitor as first line therapy
* CLL: relapsed after and/or refractory to at least two (2) prior lines of therapy. Participants with CLL are not required to have had therapy containing anti-CD20.

NOTE: Participants with CLL may be eligible after one (1) prior line of therapy if they have either:

* 17p deletion
* TP53 mutation or deletion
* Received both a Bruton's Tyrosine Kinase (BTK) inhibitor AND a B-cell lymphoma 2 (BCL2) inhibitor as first line therapy

NOTE: Participants must not have received prior treatment with a cluster of differentiation 47 (CD47) or signal regulatory protein (SIRP) targeting agent

-Adequate tissue from diagnostic biopsy (archival or fresh) must be available for performance of correlative studies

NOTE: Tumor tissue may be from any previously collected tissue and adequacy is at the discretion of the Principal Investigator. If prior tissue is not available, patient must be willing to undergo baseline tissue biopsy (for patients with known or suspected bone marrow involvement, bone marrow may be acceptable tissue per discretion of the investigator).

-Patients must have at least evaluable disease as assessed by clinical exam (i.e., palpable lymphadenopathy, measurable skin lesions, etc.), laboratory assessment (i.e., lymphoma involvement of bone marrow or peripheral blood by morphology, cytology or flow cytometry), and/or imaging (measurable lymph nodes or masses on computed tomography (CT) or magnetic resonance imaging (MRI) and/or evaluable fludeoxyglucose-18 (FDG)-avid lesions on positron emission tomography (PET). Patients may also have measurable disease.

NOTE: Patients with known active central nervous system (CNS) lymphoma are not eligible.

- Age greater than or equal to 18 years

NOTE: Because no dosing or adverse event data are currently available on the use of magrolimab in patients <18 years of age, children are excluded from this study

* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Adequate organ function as evidenced by the following laboratory parameters:

  * Absolute neutrophil count (ANC): greater than or equal to 1,000/mm(3)
  * Platelets: greater than or equal to 50,000/mcL (transfusions permitted)
  * Hemoglobin: greater than or equal to 9 g/dL (transfusions permitted). NOTE: Patients must have required fewer than 2 units of red blood cell (RBC) transfusion in the 4 weeks prior to screening. Additional transfusions after screening and prior to enrollment are acceptable.
  * Renal function: Glomerular filtration rate (GFR) greater than or equal to 30 mL/min/1.73 m(2) as estimated by the Modification of Diet in Renal Disease (MDRD) abbreviated formula. If not on target, a 24-hour urine creatinine clearance can be used to directly measure.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT): less than or equal to 3.0 x the upper limit of normal (ULN)

NOTE: Patients with liver involvement with lymphoma less than or equal to 5.0 x ULN

-Bilirubin less than or equal to 1.5 X ULN

NOTE: Patients with Gilbert's syndrome may have a bilirubin level > 1.5 X ULN, per discretion of the investigator

-The effects of the study drugs on the developing human fetus are unknown. For this reason, women of childbearing potential (WOCBP) and men must agree to use effective contraception when sexually active. This applies for the time period between signing of the informed consent form and for the following time frames after the last dose of drug, whichever is later: 90 days after the last dose of magrolimab, 30 days after the last dose of venetoclax, and 18 months after the last dose of obinutuzumab for women and 6 months after the last dose of obinutuzumab for men. Men should refrain also from donating sperm for these same timeframes, and women must also refrain from donating eggs.

NOTE: WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal (i.e., amenorrheic for >12 months without alternative medical cause; post-menopausal status in females under 55 years of age should be confirmed with a serum follicle-stimulating hormone [FSH] level within applicable local laboratory reference range for postmenopausal women). Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control (failure rate of less than 1%), e.g., intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner and sexual abstinence. The use of condoms by male patients is required unless the female partner is permanently sterile.

* Ability of patient to understand and the willingness to sign a written informed consent document
* Patients with prior autologous or allogeneic stem cell transplantation are potentially eligible if transplanted > 6 months ago, and no active graft-vs-host disease requiring immunosuppressants.

EXCLUSION CRITERIA:

* Concomitant use of any investigational anti-lymphoma treatment
* Known primary or acquired immunodeficiency syndrome (e.g., HIV) or known infection with human T-cell leukemia virus 1 (HTLV1). NOTE: HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the study drugs. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. In the future, appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* History of hemolytic anemia or autoimmune thrombocytopenia in the 3 months prior to enrollment. Patients with positive Direct Agglutination Test (DAT) but no evidence of clinically active hemolysis are eligible.
* Hepatitis B surface antigen or hepatitis B deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) positive. NOTE: Subjects who are hepatitis B core antibody positive will need to have a negative hepatitis B virus (HBV) DNA PCR result before enrollment. Those with a positive PCR for hepatitis B are excluded.
* Pregnant or breastfeeding patients. NOTE: Pregnant women are excluded in this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drugs, breastfeeding should be discontinued.
* Requirement to continue on any of the medications that have significant potential for drug-drug interactions with the study regimen. For example, the following:

  * Use of strong cytochrome P450 (CYP3A) inhibitors 7 days prior to or at initiation of venetoclax, and during ramp-up phase is contraindicated in patients with MZL, CLL and MCL. For FL patients, use of strong CYP3A inhibitors is contraindicated 7 days prior to and during the first two weeks of venetoclax treatment.
  * Consumption of one or more of the following within 3 days prior to the first dose of any study drug:

    * Grapefruit or grapefruit products
    * Seville oranges including marmalade containing Seville oranges
    * Star fruit
* Uncontrolled intercurrent illness including, but not limited to the following that may limit interpretation of results or that could increase risk to the patient at the discretion of the investigator:

  * Active hepatitis C infection. NOTE: Subjects who are hepatitis C antibody positive will need to have a negative HCV PCR result before enrollment. Those with a positive PCR for hepatitis C are excluded.
  * Any second malignancy that requires active systemic therapy
  * Known mental or physical illness that would interfere with cooperation with the requirements of the trial or confound the results or interpretation of the results of the trial and, in the opinion of the treating investigator, would make the patient inappropriate for entry into the study
  * Known active infection, or any major infection requiring treatment with intravenous (IV) antibiotics or hospitalization within 4 weeks prior to commencement of the study treatment.
* Vaccination with a live vaccine less than or equal to 28 days prior to commencement of the study treatment.
* Inability or unwillingness to swallow a large number of tablets.
* Known hypersensitivity to any of the study medications or their excipients.
* History of inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis).
* History of malabsorption syndrome felt to be significant enough to interfere with enteral absorption at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Roschewski, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0162.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Treatment: Follicular Lymphoma Dose Expansion: Magrolimab intravenous (IV) 1 mg/kg priming dose followed by 30mg/kg loading and maintenance doses + obinutuzumab IV 1000mg combination for 2 cycles (28-days each, Cycles -2 and -1), then venetoclax will be added at target dose. Triplet combination treatment with magrolimab/obinutuzumab/venetoclax will be 6 cycles (28-days each, Cycles 1-6); further treatment will be response-adapted. Obinutuzumab administered intravenously, on Days 1, 2, 8 and 15 of Cycle 1 at doses escalating from 100mg - 1000mg then on the first day for all subsequent cycles at 1000mg for dose finding phase. For expansion phase, administered on Days 1, 2, 8 and 15 of Cycle 2 at doses escalating from 100mg - 1000mg then on the first day for all subsequent cycles at 1000mg. Venetoclax for follicular lymphoma patients in dose finding phase, administered orally at a dose of 600mg or 800mg depending on tolerance, daily, cycles 1-12. For Marginal Zone Lymphoma, Mantle Cell Lymphoma or Chronic Lymphocytic Leukemia patients in dose finding phase administered at an escalating dose from 20mg-400mg Cycle 1 on days 1-35, and at a dose of 400mg per day for Cycles 2-12. Patients in expansion phase will receive target dose established from dose finding cohorts daily for all 12 cycles. Magrolimab administered intravenously, starting at 1 mg/kg on second day of first cycle then 30mg/kg on days 8, 15 and 22 of cycle 1 and days 1 and 15 of cycles 2-12 for patients in both the dose finding and expansion phases.
- Arm 1, Cohort 1 Follicular Lymphoma Level 1: Magrolimab intravenous (IV) with a 1 mg/kg dose followed by 30mg/kg doses+obinutuzumab IV 1000mg+venetoclax 800mg by mouth combination administered to 6 patients for 6 cycles (28-days each, Cycles 1-6); further treatment with additional cycles will be response-adapted. Note: Dose-limiting toxicity (DLT) assessment of the magrolimab/obinutuzumab/venetoclax triplet will take place during Cycle 1. If =2 patients experience DLT, an additional 6 patients will be enrolled at Dose level (-1) of venetoclax 600mg with magrolimab and obinutuzumab. Obinutuzumab administered IV, on Days 1, 2, 8 and 15 of Cycle 1 at doses escalating from 100mg - 1000mg then on the 1st day for all subsequent cycles at 1000mg for dose finding phase.
- Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1: Magrolimab intravenous (IV) with a 1 mg/kg priming dose followed by 30mg/kg doses + obinutuzumab IV 1000mg + venetoclax ramp-up to target dose of 400mg over 5 weeks (35 days, Cycle 1) administered to 6 patients. Triplet combination of magrolimab + obinutuzumab + venetoclax (target dose, no ramp-up) will continue for five (5) additional cycles (28-days each, Cycles 2-6); further treatment with additional cycles will be response-adapted. If =2 patients experience DLT, an additional 6 patients will be enrolled at Dose level (-1) of venetoclax 200mg with magrolimab and obinutuzumab. Obinutuzumab administered IV, on Days 1, 2, 8 and 15 of Cycle 1 at doses escalating from 100mg - 1000mg then on the first day for all subsequent cycles at 1000mg for dose finding phase.
- Experimental Treatment: Chronic Lymphocytic Leukemia Dose Expansion: Window of magrolimab intravenous (IV) with a 1 mg/kg priming dose followed by 30mg/kg loading and maintenance doses + obinutuzumab IV 1000mg combination for two (2) cycles (28-day cycles, Cycles -2 and -1), then venetoclax safety ramp-up to target dose (dose determined from Arm 2) over 5 weeks (35-days, Cycle 1). Triplet combination treatment with magrolimab + obinutuzumab + venetoclax (target dose, no ramp-up) will continue for 5 additional cycles (28-days each, Cycles 2-6); further treatment will be response-adapted. Obinutuzumab administered intravenously, on Days 1, 2, 8 and 15 of Cycle 1 at doses escalating from 100mg - 1000mg then on the first day for all subsequent cycles at 1000mg for dose finding phase.
Period: Overall Study
Arm/Group | Experimental Treatment: Follicular Lymphoma Dose Expansion | Arm 1, Cohort 1 Follicular Lymphoma Level 1 | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1 | Experimental Treatment: Chronic Lymphocytic Leukemia Dose Expansion
Started | 0 | 5 | 6 | 0
Off Study- Study is Cancelled | 0 | 5 | 6 | 0
Completed | 0 | 5 | 4 | 0
Not Completed | 0 | 0 | 2 | 0
Not completed — Dose limiting toxicity | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1, Cohort 1 Follicular Lymphoma Level 1 | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1 | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (13.5) | 69.17 (7.14) | 64.27 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 0 | 3 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Grades 3, 4, and/or 5 Dose-limiting Toxicities (DLT) Probably and/or Definitely Related to Triplet Combination Therapy
Description: Incidence of dose limiting toxicities (i.e., grade and frequency) to determine safety and tolerability were measured by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade is 3 is severe. Grade 4 is life threatening, and Grade 5 is death related to adverse event. A DLT is defined as any grade 3 or higher adverse event that is clinically relevant and deemed probably or definitely related to any of the study drugs or to the combination therapy and occurs during the venetoclax dose-finding period. Exceptions are non-hematologic grade 3 nausea, vomiting or diarrhea. Grade 3 fatigue, electrolyte disturbances, magrolimab or obinutuzumab infusion reactions, and/or grade 3 laboratory abnormalities. Hematologic grade 3 neutropenia, thrombocytopenia, anemia and hemolytic anemia. And/or grade 3 or 4 lymphopenia.
Time Frame: 4 weeks for Arm 1 and 5 weeks for Arm 2
Measure: Number; unit: Adverse events
Arm/Group | Arm 1, Cohort 1 Follicular Lymphoma Level 1 | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1
Number analyzed (Participants) | 5 | 6
Adverse events
  Grade 4 Thrombocytopenia Definitely Related | 0 | 2
  Grade 3 and 5 Probably and/or Definitely Related Toxicity | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR) (Complete Response + Partial Response)
Description: ORR was determined and reported from individual cohorts and histological diagnosis. ORR was measured by the Lugano response criteria for Follicular Lymphoma, Mantle Cell Lymphoma and Marginal Zone Lymphoma; and the International Workshop on Chronic Lymphocytic Leukemia criteria for Chronic Lymphocytic Leukemia. Complete response is complete resolution of the lesion on imaging. Partial response is 50% or greater reduction in the maximum diameter of the lesion from its original tumor size on imaging. Disease progression is an increase of 50% or more in size of a previously involved site measuring ≥1.5 cm.
Time Frame: From the start of the treatment until disease progression/recurrence, median follow-up of 17.4 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1, Cohort 1 Follicular Lymphoma Level 1 | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1
Number analyzed (Participants) | 5 | 6
Percentage of participants
  Complete Response | 40 [7.1 to 76.9] | 66.7 [30.0 to 94.1]
  Partial Response | 40 [7.1 to 76.9] | 16.7 [0.9 to 56.4]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was estimated using Kaplan-Meier curves and reported along with a 95% confidence interval. DOR was measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, death, or, in the absence of progressive disease (PD), date of last assessment. DOR was measured by the Lugano response criteria for Follicular Lymphoma, Mantle Cell Lymphoma and Marginal Zone Lymphoma; and the International Workshop on Chronic Lymphocytic Leukemia criteria for Chronic Lymphocytic Leukemia. Complete response is complete resolution of the lesion on imaging. Partial response is 50% or greater reduction in the maximum diameter of the lesion from its original tumor size on imaging. Disease progression is an increase of 50% or more in size of a previously involved site measuring ≥1.5 cm.
Time Frame: From the start of the treatment until time of disease relapse, disease progression, or death, whichever occurs first, an average of 10.9 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1, Cohort 1 Follicular Lymphoma Level 1 | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1
Number analyzed (Participants) | 5 | 6
Months | 17.5 [2.8 to NA] — Upper confidence interval was not reached | NA [NA to NA] — Median and 95% confidence interval cannot be calculated because it was not reached.

4. Secondary Outcome: Event-free Survival (EFS)
Description: EFS was estimated using Kaplan-Meier curves and reported along with a 95% confidence interval. EFS is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, alternative anti-lymphoma therapy including radiation, or death, whichever occurs first, measured by the Lugano response criteria for Follicular Lymphoma, Mantle Cell Lymphoma and Marginal Zone Lymphoma; and the International Workshop on Chronic Lymphocytic Leukemia criteria for Chronic Lymphocytic Leukemia. Disease progression is an increase of 50% or more in size of a previously involved site measuring ≥1.5 cm.
Time Frame: From the start of the treatment until time of disease relapse, disease progression, alternative anti-lymphoma therapy including radiation, or death, whichever occurs first, up to 20 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1, Cohort 1 Follicular Lymphoma Level 1 | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1
Number analyzed (Participants) | 5 | 6
Months | 20.0 [1.5 to NA] — Upper confidence interval was not reached. | NA [NA to NA] — Median and 95% confidence interval cannot be calculated because it was not reached.

5. Secondary Outcome: Progression-free Survival
Description: PFS was estimated using Kaplan-Meier curves and reported along with a 95% confidence interval. PFS is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, or death, whichever occurs first. PFS was measured by the Lugano response criteria for Follicular Lymphoma, Mantle Cell Lymphoma and Marginal Zone Lymphoma; and the International Workshop on Chronic Lymphocytic Leukemia criteria for Chronic Lymphocytic Leukemia. Disease progression is an increase of 50% or more in size of a previously involved site measuring ≥1.5 cm.
Time Frame: From the start of the treatment until time of disease relapse, disease progression, or death, whichever occurs first, an average of 13.9 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1, Cohort 1 Follicular Lymphoma Level 1 | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1
Number analyzed (Participants) | 5 | 6
Months | 20.2 [1.5 to NA] — Upper confidence interval was not reached. | NA [NA to NA] — Median and 95% confidence interval cannot be calculated because it was not reached.

6. Secondary Outcome: Overall Survival (OS)
Description: OS was estimated using Kaplan-Meier curves and reported along with a 95% confidence interval. OS is defined as the time from study enrollment until death from any cause.
Time Frame: From the start of the treatment until death from any cause, an average of 15.6 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1, Cohort 1 Follicular Lymphoma Level 1 | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1
Number analyzed (Participants) | 5 | 6
Months | NA [NA to NA] — Median and 95% confidence interval cannot be calculated because it was not reached because of insufficient number of participants with events (i.e., deaths). | NA [NA to NA] — Median and 95% confidence interval cannot be calculated because it was not reached because of insufficient number of participants with events (i.e., deaths).

7. Secondary Outcome: Percentage of Participants With Chronic Lymphocytic Leukemia (CLL) With Complete Molecular Remission (MRD Negativity)
Description: The percentage of participants who are MRD negative was determined by circulating tumor deoxyribonucleic acid (ctDNA) assay after therapy. Negative is undetectable CLL cells on peripheral blood flow cytometry after end of treatment.
Time Frame: From the start of the treatment until disease progression/recurrence, an average of 3.3 months.
Population: This outcome measure is applicable to participants with CLL only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1
Number analyzed (Participants) | 6
percentage of participants | 100 [18 to 100]

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From the first study intervention, Day 1 through 30 days after the last dose of study agent was administered, an average of 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Cohort 1 Follicular Lymphoma Level 1 | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1
Number analyzed (Participants) | 5 | 6
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: All-Cause Mortality monitored/assessed an average of 15.6 months, Adverse Events monitored/assessed from Day 1 through 30 days after the last dose of study agent was administered, an average of 6 months.
Arm/Group | Arm 1, Cohort 1 Follicular Lymphoma Level 1 | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/6
Other Adverse Events (participants affected / at risk) | 5/5 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, Cohort 1 Follicular Lymphoma Level 1 (N=5) | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1 (N=6)
Lung infection (Infections and infestations) | 1 (2) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, Cohort 1 Follicular Lymphoma Level 1 (N=5) | Arm 2, Cohort 2 Marginal Zone Lymphoma, Mantle Cell Lymphoma, & Chronic Lymphocytic Leukemia Level 1 (N=6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, SARS-COV-2 (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lung infection (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (4)
Platelet count decreased (Investigations) | 2 (5) | 2 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT04599634/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Screening Consent, Affected Patient (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT04599634/ICF_001.pdf
  • Informed Consent Form: Cohort Affected Patient Consent (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT04599634/ICF_002.pdf